CLINICAL TRIAL: NCT02299050
Title: Effect of Cycloset on Glycemic Control in Type 2 Diabetic Patients Inadequately Controlled on GLP-1 Analogue Therapy
Brief Title: Effect of Cycloset on Glycemic Control When Added to Glucagon-like Peptide 1 (GLP-1) Analogue Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: VeroScience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20130330H
Record Dates: First submitted 2014-09-16; First posted 2014-11-24 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; T2DM; Cycloset; Glycemic Control; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cycloset (Other): Drug - Cycloset Cycloset 2.4 -3.2 mg/day
  Other Names:
  Bromocriptine Mesylate Quick Release
  Interventions: Drug: Cycloset

INTERVENTIONS:
Drug: Cycloset — Bromocriptine QR 0.8 mg tablet 0.8 mg/day with dose increased to a maximum of 3.2 mg/day or as tolerated to a minimum of 2.4 mg/day Other names: Cycloset, B-QR
  Other Names: Bromocriptine Mesylate Quick Release

SUMMARY:
Purpose This study will examine the effect of the addition of Cycloset upon glucose metabolism (glycemic control including post prandial glucose metabolism) in individuals with inadequately controlled (HbA1c 7.5-10.0) type 2 diabetes (T2DM) who are already on Bydureon (exenatide once weekly) or Victoza (liraglutide once daily) as part of their standard care.

Both a mechanistic rationale and empirical experimental evidence implicate a beneficial interaction between bromocriptine and the incretin mimetics (GLP-1 analogs) upon postprandial hyperglycemia in insulin resistant states. One of the actions of the incretin mimetics such as the GLP-1 analogs is to stimulate postprandial beta cell insulin secretory response to plasma glucose (see drug labeling information; www.fda.gov). Thus the combination of Cycloset that is working as a post prandial insulin sensitizier with therapies that increase post prandial insulin would be expected to provide complimentary glucose lowering effects. To date, however, no such studies investigating the interactive effects of a GLP-1 analog and Bromocriptine-QR (QR=extended release) (Cycloset) have been conducted in humans.

Condition - Type 2 Diabetes. Intervention - Cycloset. Phase - Phase 4

Study Type: Interventional Study Design: Treatment, Single Group Assignment, Open Label, N/A, Safety/Efficacy Study

Official Title: Effect of Cycloset on Glycemic Control in Type 2 Diabetic Patients Inadequately Controlled on GLP-1 Analogue Therapy

DETAILED DESCRIPTION:
This is a single-site, prospective, cohort study that will assess the effect of Cycloset as add-on therapy in adult subjects with T2DM that is inadequately controlled (HbA1c 7.5% to 10.0%) on GLP-1 analog therapy with either exenatide (Bydureon) once weekly or liraglutide (Victoza) once daily.

Entry criteria will be checked at the screening visit. All qualified subjects will undergo baseline studies including non-invasive hemodynamic testing for assessment of aortic stiffness and pulse wave velocity, assessment of body weight composition by dual-energy X-ray absorptiometry (DXA), assessment of endothelial function using the Endo-PAT device, measurement of cytokines and inflammatory biomarkers in the peripheral blood and urine, assessment of oxidative stress and inflammatory markers in white blood cells isolated from a peripheral whole blood sample, a 5-hour mixed meal tolerance test (MMT) for assessment of postprandial glucose metabolism and 24-hour ambulatory BP monitoring.

Following completion of all the baseline studies as above, subjects will be started on Cycloset, 0.8 mg/day in addition to their stable dose of Bydureon (exenatide) (2mg/week) or Victoza (liraglutide) (1.2-1.8 mg/day), and the dose will be increased by 0.8 mg/day every week to a maximum of 3.2 mg/day, or as tolerated to a minimum of 2.4 mg/day.

Subjects will return at months 1, 2, 3, and 4 for interim medical history, body weight, HbA1c, and FPG (Fasting plasma glucose). Postural blood pressure measurements will be obtained with the subject lying down and then after standing for 5 minutes at each of the visits. At month 4, all of the baseline studies detailed above will be repeated.

All tests will be performed in the Clinical Research Center at the Texas Diabetes Institute/University of Texas Health Science Center, San Antonio.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes male or female subjects between the ages of 30 and 70 years of age, inclusive, at Screening
* BMI = 24-40 kg/m2
* HbA1c = 7.5-10.0%
* Stable body weight (±3-4lbs) over the preceding 3 months
* Subjects currently receiving a stable dose of exenatide (2mg/week) or liraglutide (1.2-1.8 mg/day) for at least 90 days prior to determination of baseline HbA1C and eligibility for enrollment in the study protocol.
* Subjects with a daytime feeding/night time sleeping schedule
* Subjects with no evidence of major organ system disease as determined by physical exam, history, and screening laboratory data
* Women must be of non-childbearing potential as defined by one of the following:
* Women >45 and < 60 years of age at Screening, who have been amenorrheic for at least 2 years
* Women who have had a documented hysterectomy and/or bilateral oophorectomy
* Women > 60 years of age
* Females of childbearing potential with a negative pregnancy test at Screening and Treatment visits, using one of the following forms of contraception for the duration of participation in the study (i.e., until Follow-up 7-14 days post last dose): Oral contraceptive, Injectable progesterone, subdermal implant, spermicidal foam/gel/film/cream/suppository, diaphragm with spermicide, copper or hormonal containing IUD (intrauterine device), sterile male partner vasectomized > 6 month pre-dosing
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Subjects must be willing and able to comply with scheduled visits, treatment, laboratory tests and study procedures.

Exclusion Criteria:

* Recent (i.e., within three (3) months prior to Screening) evidence or medical history of unstable concurrent disease such as: documented evidence or history of clinically significant hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, immunological, or clinically significant neurological disease.
* No history of T2DM
* BMI of less 24 and greater 40 kg/m2
* Unstable body weight (change of greater than ±3-4lbs over the preceding 3 months
* Subjects not currently receiving exenatide or liraglutide
* Subjects participating in an excessively heavy exercise program
* Subject with a feeding/sleeping schedule different from a daytime feeding/night time sleeping schedule
* Subjects taking medications known to alter glucose metabolism (with the exception of metformin and/or pioglitazone) or which effect brain neuro synaptic function are excluded.
* Subjects with evidence of major organ system disease as determined by physical exam, history, and screening laboratory data
* Pregnant subjects or subjects unwilling to use birth control during their study enrollment
* Blood donation of approximately 1 pint (500 mL) within 8 weeks prior to Screening 12. Subjects that are allergic to bromocriptine or any of the other ingredients in Cycloset, or take ergot medicines, breastfeeding or have history of syncope or Type 1 diabetes mellitus
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results that, in the judgment of the investigator, would make the subject inappropriate for entry into this study subjects of reproductive potential

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-06; Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cycloset: Drug - Cycloset Cycloset 2.4 -3.2 mg/day
  Other Names:
  Bromocriptine Mesylate Quick Release
  Cycloset: Bromocriptine QR 0.8 mg tablet 0.8 mg/day with dose increased to a maximum of 3.2 mg/day or as tolerated to a minimum of 2.4 mg/day Other names: Cycloset, B-QR
Period: Overall Study
Arm/Group | Cycloset
Started | 23
Completed | 15
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: Subjects who were consented and received study intervention
Arm/Group | Cycloset
Number analyzed (Participants) | 15
Age, Customized [Mean (Standard Deviation); unit: years]
  Participants age | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
Region of Enrollment [Number; unit: participants]
  United States | 15
Medications currently used for type 2 diabetes [Count of Participants; unit: Participants]
  Liraglutide (1.2 - 1.8 mg/d) | 15
  Metformin | 12
  Low dose glargine insulin | 3

OUTCOME MEASURES:

1. Primary Outcome: HbA1C
Description: The objective of this study is to examine the effect of the addition of Cycloset on glycemic control in inadequately controlled (HbA1c 7.5-10.0) T2DM (type 2 diabetes mellitus) patients who are already on Bydureon (exenatide once weekly) or Victoza (liraglutide ) as part of their standard care.
  An additional co-primary objective of the study is to examine the effect of Cycloset on postprandial glucose metabolism.
Time Frame: Change from baseline to four to five months
Measure: Mean (Standard Error); unit: mmol/mol
Arm/Group | Cycloset
Number analyzed (Participants) | 15
mmol/mol
  Baseline Measurement | 8.3 (0.3)
  Measurement at 4-5 months | 7.7 (0.2)

2. Primary Outcome: Glucose Metabolism During Mixed Meal Tolerance Test
Description: The objective of this study is to examine the effect of the addition of Cycloset on glycemic control in inadequately controlled (HbA1c 7.5-10.0) T2DM patients who are already on Bydureon (exenatide once weekly) or Victoza (liraglutide ) as part of their standard care.
Time Frame: Change from baseline to four to five months
Measure: Mean (Standard Error); unit: mg/kg *min
Arm/Group | Cycloset
Number analyzed (Participants) | 15
mg/kg *min
  Baseline Measurement | 1.1 (0.1)
  Measurement at 4-5 months | 0.7 (0.1)

3. Secondary Outcome: Endothelial Function,
Description: To assess the potential beneficial effect of Cycloset on endothelial function. This is measured by using pulse pressure.
Time Frame: Change from baseline to four to five months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Cycloset
Number analyzed (Participants) | 15
mmHg
  Baseline Measurement | 54 (2)
  Measurement at 4-5 months | 51 (2)

4. Secondary Outcome: Body Composition
Description: To assess the potential beneficial effect of Cycloset on body weight composition.
Time Frame: Change from baseline to four to five months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Cycloset
Number analyzed (Participants) | 15
kg
  Baseline Measurement | 88.1 (13.8)
  Measurement at 4-5 months | 87.1 (13.7)

5. Secondary Outcome: Percentage Body Fat
Description: To assess the potential beneficial effect of Cycloset on body fat content
Time Frame: Change from baseline to four to five months
Measure: Mean (Standard Error); unit: percentage body fat
Arm/Group | Cycloset
Number analyzed (Participants) | 15
percentage body fat
  Baseline Measurement | 39.1 (6.7)
  Measurement at 4-5 months | 39.3 (7.4)

6. Secondary Outcome: Blood Pressure
Description: To assess the potential beneficial effect of Cycloset on blood pressure.
Time Frame: Change from baseline to four to five months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Cycloset
Number analyzed (Participants) | 15
mmHg
  Systolic pressure at baseline | 134 (4)
  Systolic pressure at 4-5 months | 126 (6)
  Diastolic pressure at baseline | 78 (3)
  Diastolic pressure at 4-5 months | 73 (4)

7. Secondary Outcome: Mean Arterial Blood Pressure
Description: To assess the potential beneficial effect of Cycloset on change in mean arterial blood pressure
Time Frame: Change from baseline to four to five months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Cycloset
Number analyzed (Participants) | 15
mmHg
  Baseline Measurement | 97 (5)
  Measurement at 4-5 months | 90 (4)

8. Secondary Outcome: Arterial Stiffness (AS)
Description: To assess the potential beneficial effect of Cycloset on arterial stiffness. Arterial stiffness is calculated by the measurement of pulse pressure, where Pulse pressure = SBP - DBP (Where SBP is systolic blood pressure and DBP is diastolic blood pressure) The calculated value is used as a predictor of cardiovascular disease. Higher values indicate that cardiovascular disease is more likely.
Time Frame: Change from baseline to four to five months
Measure: Mean (Standard Error); unit: au (arbitrary units)
Arm/Group | Cycloset
Number analyzed (Participants) | 15
au (arbitrary units)
  Baseline Measurement | 19.8 (4.1)
  Measurement at 4-5 months | 16.2 (3.7)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from baseline to between 4 to 5 months
Arm/Group | Cycloset
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycloset (N=15)
Orthostatic Hypotension (Cardiac disorders) | 2 (2) — Low blood pressure when standing up too quickly
Light-headedness (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT02299050/Prot_SAP_000.pdf